CLINICAL TRIAL: NCT03838237
Title: Effect of Migalastat on Cardiac Involvement in Fabry Disease
Acronym: MAIORA
Status: Completed | Type: Observational
Sponsor: Ospedale San Donato (Other)
Collaborators: Amicus Therapeutics (Industry); Institute of Biomedicine and Molecular Immunology - CNR (Unknown)
Responsible Party: Principal Investigator, Antonia Camporeale, MD, PhD, Ospedale San Donato
Other Study IDs: 148/int/2017
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Fabry Disease; Heart Diseases
Keywords: Fabry Disease; Migalastat; Cardiomyopathy; Cardiac Magnetic Resonance; T1 mapping
MeSH Terms: conditions — Fabry Disease; Heart Diseases; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for Troponin T, NT-proBNP and microRNA assay
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry Disease patients: Patients with genetic diagnosis of Fabry Disease, clinical indication to Migalastat and signs of cardiac involvement (early or advanced) will undergo cardiological evaluation before and 18 months after therapy with Migalastat (123 mg every other day)
  Interventions: Diagnostic Test: Cardiological evaluation

INTERVENTIONS:
Diagnostic Test: Cardiological evaluation — Baseline evaluation
  * FAbry STabilization indEX (FASTEX)
  * 12 leads ECG
  * Blood samples for microRNA, TnT HS and NT-proBNP dosages
  * 2D echocardiogram
  * Cardio-pulmonary test
  * Contrast-enhanced CMR including:
    * Cine images
    * T2 mapping sequences
    * T1 mapping sequences before and 15' after contrast medium administration
    * Late Gadolinium Enhancement (LGE) imaging
    * Phase contrast images (LVOT, aortic flow)
  Follow up evaluation
  •After 18 months, the same procedures will be repeated

SUMMARY:
Anderson-Fabry Disease (AFD) is one of the rare lysosomal storage disorders for which a cause - specific therapy is available. Recently, a new specific drug has been marketed, namely Migalastat, a small-molecule pharmacological chaperone. The effect of Migalastat on cardiac involvement has been assessed so far by 2D echocardiography, demonstrating a significant reduction in left ventricular (LV) mass after 18 months of therapy. Calculation of LV mass by 2D echocardiography is limited by geometrical assumptions and quality of echocardiographic window, with a strong impact on accuracy. Cardiac Magnetic Resonance (CMR) overcomes these limitations, thus representing the gold standard technique for ventricular mass, volumes and function estimation. Moreover, CMR offers the unique possibility to perform a non-invasive tissue characterization, including the detection of both myocardial fibrosis by Late Gadolinium Enhancement and sphingolipid storage by T1 mapping. Beyond an accurate morphological description and a detailed tissue characterization, a complete cardiological assessment should also integrate functional data and bio-humoral profile.

This study is designed to provide a comprehensive evaluation of the therapeutic effect of Migalastat (123 mg every other day) on cardiac involvement after 18 months of therapy, integrating a morphological, functional and bio-humoral assessment.

DETAILED DESCRIPTION:
Anderson-Fabry disease is a rare X-linked lysosomal disorder, mainly affecting cardiovascular, renal and nervous systems. Cardiac injury is the leading cause of death in these patients. Heart involvement is characterized by left ventricular hypertrophy (LVH), myocardial scarring and/or inflammation, Bradyarrhythmias or tachyarrhythmias, heart failure and represents the main cause of death in these patients. Since 2001, specific therapies (enzyme replacement therapy (ERT) first and pharmacological chaperone migalastat more recently) are available to treat these patients.

Migalastat is a small-molecule pharmacological chaperone stabilizing speciﬁc mutant forms of the enzyme (α-Gal ) and promoting its catabolic function. These mutant forms of α-Gal are deﬁned as amenable to Migalastat. In patients with amenable mutations, orally administered Migalastat is a potential alternative treatment to intravenous ERT. Because of its chemical nature (small molecule) and route of administration (orally), Migalastat would avoid ERT-associated immunogenicity and infusion-associated reactions. Additionally, the higher volume of distribution of migalastat relative to ERT suggests enhanced penetration of organs and tissues. Theoretically, the chaperoning of α-Gal by Migalastat to lysosomes may better mimic natural enzyme trafficking and result in more constant α-Gal activity than biweekly ERT infusions.

Two main clinical studies have been published so far about safety and efficacy of Migalastat in AFD, demonstrating good safety, tolerability and comparable efficacy to ERT. These studies reported a significant decrease in LV mass index assessed by 2D echocardiography (-6,6 g/m2 in 33 patients after 18 months of therapy), mostly in patients with overt cardiac involvement and greater than the changes observed with ERT (-2 g/m2 in 16 patients after 18 months of therapy).

Calculation of LV mass by 2D echocardiography is based on the "Devereux formula", assuming that the LV is a prolate ellipsoid with a 2:1 long/short axis ratio and symmetric distribution of hypertrophy. This is not always the case in AFD Cardiomyopathy, showing a wide variety of hypertrophy patterns. Moreover, since linear measurements of LV wall thickness and diameters are cubed in this formula, even small measurement errors in dimensions or thickness have a strong impact on accuracy.

Cardiac magnetic resonance (CMR) represents the gold standard technique for ventricular mass, volumes and function estimation because of the possibility to directly measure these parameters without geometrical assumption. Therefore, CMR has an excellent inter-study reproducibility both in normal and in pathologic hearts, overcoming 2D echocardiography. Beyond its high reproducibility in LV mass measurement, CMR offers the unique possibility of non-invasive tissue characterization. This concept includes both detection and quantification of myocardial fibrosis by Late Gadolinium Enhancement images and application of new techniques, namely T1 mapping, detecting myocardial sphingolipid storage even before LVH occurs. Also, CMR allows a detailed characterization of myocardial deformation by feature tracking. Feature tracking CMR (FT-CMR) approximately applies the same principles of speckle tracking echocardiography (even though with differences methods of image acquisition and reconstruction) in order to measure global and segmental myocardial deformation. The strength of FT-CMR consists of its relatively unrestricted access to large fields of view, its high spatial resolution and its relatively high signal to noise and contrast to noise ratios.

MicroRNAs (miRNAs) are small noncoding RNAs that regulate gene expression at the post-transcriptional level. MiRNAs have emerged as key regulators of several physiological and pathophysiological processes. Besides their intracellular function, recent studies demonstrated that miRNAs can be exported or released by cells and circulate in blood in a remarkably stable form. The discovery of circulating miRNAs opens the possibilities to use circulating miRNA patterns as biomarkers for several pathologies also for cardiovascular diseases. In a recent study, a common microRNA signature in AFD patients regardless of gender and age has been identified.15 miRNAs differentially expressed between 10 AFD subjects and 10 normal controls (NC) have been found. The levels of these 15 miRNAs in plasma sample of 10 subjects with LVH and no mutation in the Galactosidase Alpha (GLA) gene have also been studied. Among these 15 miRNAs, 3 discriminated AFD patients from subjects with LVH. In particular, 2 microRNAs (mir-199a-5p and mir126a-3p) were up-regulated and 1 miRNA (mir-423-5p) was down-expressed in AFD patients. Interestingly, in a recent study increased plasmatic levels of miR-126 and miR-199a were significantly associated with a lower major adverse Cardiovascular (CV) event rate in patients with coronary artery disease. Instead, elevated plasmatic levels of mir-423-5p is strongly related to the clinical diagnosis of Heart Failure. Several evidences indicate that the aberrantly expressed plasmatic miRNAs in AFD are linked to microvascular or macrovascular damage involved in the typical AFD vasculopathy and could be attractive as diagnostic markers as well as for the monitoring of the pharmacological treatment.

Integration of all these aspects allows a complete morpho-functional evaluation of cardiac involvement in AFD and a detailed monitoring of the effects of specific drugs.

This study is designed to provide a comprehensive evaluation of the therapeutic effect of Migalastat on cardiac involvement, integrating a morphological, functional and bio-humoral assessment of heart involvement. 15 patients with amenable mutation, clinical indication to Migalastat and signs of early or overt cardiac involvement with will undergo a complete cardiological evaluation before and 18 months after therapy with Migalastat. The cardiological assessment will include ECG, 2D echocardiography, CMR, cardio-pulmonary test, dosage of peripheral biomarkers (TnT High Sensitive; NT-proBNP, mir-199a-5p and mir126a-3p, mir-423-5p).

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Fabry Disease and amenable mutation
* Clinical indication to Migalastat
* Signs of clinical or preclinical cardiac involvement (low T1 values with or without left ventricular hypertrophy)
* Age >16
* Ability to give a complete informed consent (for minor patients informed consent will be given by parents)

Exclusion Criteria:

* Contraindication to Migalastat (pregnancy, age <16, Glomerular Filtration Rate <30 ml/min, hypersensitivity to the active ingredient)
* Contraindication to CMR study (metallic fragment or foreign body, known claustrophobia, PaceMaker/Implantable Cardioverter Defibrillator not CMR conditional, electronic implant or device, eg, insulin pump or other infusion pump)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between patients with genetic diagnosis of AFD referred for CMR at Policlinico San Donato, 15 patients with amenable mutation, clinical indication to Migalastat and signs of early or overt cardiac involvement (low myocardial native T1 value ± left ventricular hypertrophy) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Delta left ventricular mass | 18 months
  Changes in left ventricular mass measured by cardiac magnetic resonance

SECONDARY OUTCOMES:
Delta native myocardial T1 values | 18 months
  Changes in native myocardial T1 values measured by cardiac magnetic resonance
Delta left ventricular global longitudinal strain | 18 months
  Changes in left ventricular global longitudinal strain measured by cardiac magnetic resonance
Delta 3 plasmatic microRNAs levels | 18 months
  Changes in mir-199a-5p, mir126a-3p, mir-423-5p levels measured by Real-Time quantitative Polymerase Cycle Reaction (RT-qPCR)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Camporeale, MD, PhD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

REFERENCES:
- [Background] Hughes DA, Nicholls K, Shankar SP, Sunder-Plassmann G, Koeller D, Nedd K, Vockley G, Hamazaki T, Lachmann R, Ohashi T, Olivotto I, Sakai N, Deegan P, Dimmock D, Eyskens F, Germain DP, Goker-Alpan O, Hachulla E, Jovanovic A, Lourenco CM, Narita I, Thomas M, Wilcox WR, Bichet DG, Schiffmann R, Ludington E, Viereck C, Kirk J, Yu J, Johnson F, Boudes P, Benjamin ER, Lockhart DJ, Barlow C, Skuban N, Castelli JP, Barth J, Feldt-Rasmussen U. Oral pharmacological chaperone migalastat compared with enzyme replacement therapy in Fabry disease: 18-month results from the randomised phase III ATTRACT study. J Med Genet. 2017 Apr;54(4):288-296. doi: 10.1136/jmedgenet-2016-104178. Epub 2016 Nov 10. PMID 27834756
- [Background] Sado DM, White SK, Piechnik SK, Banypersad SM, Treibel T, Captur G, Fontana M, Maestrini V, Flett AS, Robson MD, Lachmann RH, Murphy E, Mehta A, Hughes D, Neubauer S, Elliott PM, Moon JC. Identification and assessment of Anderson-Fabry disease by cardiovascular magnetic resonance noncontrast myocardial T1 mapping. Circ Cardiovasc Imaging. 2013 May 1;6(3):392-8. doi: 10.1161/CIRCIMAGING.112.000070. Epub 2013 Apr 5. PMID 23564562
- [Background] Patel V, O'Mahony C, Hughes D, Rahman MS, Coats C, Murphy E, Lachmann R, Mehta A, Elliott PM. Clinical and genetic predictors of major cardiac events in patients with Anderson-Fabry Disease. Heart. 2015 Jun;101(12):961-6. doi: 10.1136/heartjnl-2014-306782. Epub 2015 Feb 5. PMID 25655062
- [Background] Linhart A, Elliott PM. The heart in Anderson-Fabry disease and other lysosomal storage disorders. Heart. 2007 Apr;93(4):528-35. doi: 10.1136/hrt.2005.063818. No abstract available. PMID 17401074
- [Background] Moon JC, Sheppard M, Reed E, Lee P, Elliott PM, Pennell DJ. The histological basis of late gadolinium enhancement cardiovascular magnetic resonance in a patient with Anderson-Fabry disease. J Cardiovasc Magn Reson. 2006;8(3):479-82. doi: 10.1080/10976640600605002. PMID 16755835
- [Background] Eng CM, Guffon N, Wilcox WR, Germain DP, Lee P, Waldek S, Caplan L, Linthorst GE, Desnick RJ; International Collaborative Fabry Disease Study Group. Safety and efficacy of recombinant human alpha-galactosidase A replacement therapy in Fabry's disease. N Engl J Med. 2001 Jul 5;345(1):9-16. doi: 10.1056/NEJM200107053450102. PMID 11439963
- [Background] Schiffmann R, Kopp JB, Austin HA 3rd, Sabnis S, Moore DF, Weibel T, Balow JE, Brady RO. Enzyme replacement therapy in Fabry disease: a randomized controlled trial. JAMA. 2001 Jun 6;285(21):2743-9. doi: 10.1001/jama.285.21.2743. PMID 11386930
- [Background] Weidemann F, Breunig F, Beer M, Sandstede J, Turschner O, Voelker W, Ertl G, Knoll A, Wanner C, Strotmann JM. Improvement of cardiac function during enzyme replacement therapy in patients with Fabry disease: a prospective strain rate imaging study. Circulation. 2003 Sep 16;108(11):1299-301. doi: 10.1161/01.CIR.0000091253.71282.04. Epub 2003 Sep 2. PMID 12952834
- [Background] Imbriaco M, Pisani A, Spinelli L, Cuocolo A, Messalli G, Capuano E, Marmo M, Liuzzi R, Visciano B, Cianciaruso B, Salvatore M. Effects of enzyme-replacement therapy in patients with Anderson-Fabry disease: a prospective long-term cardiac magnetic resonance imaging study. Heart. 2009 Jul;95(13):1103-7. doi: 10.1136/hrt.2008.162800. Epub 2009 Apr 15. PMID 19372091
- [Background] Germain DP, Weidemann F, Abiose A, Patel MR, Cizmarik M, Cole JA, Beitner-Johnson D, Benistan K, Cabrera G, Charrow J, Kantola I, Linhart A, Nicholls K, Niemann M, Scott CR, Sims K, Waldek S, Warnock DG, Strotmann J; Fabry Registry. Analysis of left ventricular mass in untreated men and in men treated with agalsidase-beta: data from the Fabry Registry. Genet Med. 2013 Dec;15(12):958-65. doi: 10.1038/gim.2013.53. Epub 2013 May 23. PMID 23703683
- [Background] Beer M, Weidemann F, Breunig F, Knoll A, Koeppe S, Machann W, Hahn D, Wanner C, Strotmann J, Sandstede J. Impact of enzyme replacement therapy on cardiac morphology and function and late enhancement in Fabry's cardiomyopathy. Am J Cardiol. 2006 May 15;97(10):1515-8. doi: 10.1016/j.amjcard.2005.11.087. Epub 2006 Mar 29. PMID 16679096
- [Background] Germain DP, Charrow J, Desnick RJ, Guffon N, Kempf J, Lachmann RH, Lemay R, Linthorst GE, Packman S, Scott CR, Waldek S, Warnock DG, Weinreb NJ, Wilcox WR. Ten-year outcome of enzyme replacement therapy with agalsidase beta in patients with Fabry disease. J Med Genet. 2015 May;52(5):353-8. doi: 10.1136/jmedgenet-2014-102797. Epub 2015 Mar 20. PMID 25795794
- [Background] Germain DP, Fan JQ. Pharmacological chaperone therapy by active-site-specific chaperones in Fabry disease: in vitro and preclinical studies. Int J Clin Pharmacol Ther. 2009;47 Suppl 1:S111-7. PMID 20040321
- [Background] Johnson FK, Mudd PN Jr, Bragat A, Adera M, Boudes P. Pharmacokinetics and Safety of Migalastat HCl and Effects on Agalsidase Activity in Healthy Volunteers. Clin Pharmacol Drug Dev. 2013 Apr;2(2):120-32. doi: 10.1002/cpdd.1. Epub 2013 Feb 21. PMID 27121667
- [Background] Khanna R, Soska R, Lun Y, Feng J, Frascella M, Young B, Brignol N, Pellegrino L, Sitaraman SA, Desnick RJ, Benjamin ER, Lockhart DJ, Valenzano KJ. The pharmacological chaperone 1-deoxygalactonojirimycin reduces tissue globotriaosylceramide levels in a mouse model of Fabry disease. Mol Ther. 2010 Jan;18(1):23-33. doi: 10.1038/mt.2009.220. Epub 2009 Sep 22. PMID 19773742
- [Background] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Deva DP, Hanneman K, Li Q, Ng MY, Wasim S, Morel C, Iwanochko RM, Thavendiranathan P, Crean AM. Cardiovascular magnetic resonance demonstration of the spectrum of morphological phenotypes and patterns of myocardial scarring in Anderson-Fabry disease. J Cardiovasc Magn Reson. 2016 Mar 31;18:14. doi: 10.1186/s12968-016-0233-6. PMID 27036375
- [Background] Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol. 2002 Jul 1;90(1):29-34. doi: 10.1016/s0002-9149(02)02381-0. PMID 12088775
- [Background] Moon JC, Sachdev B, Elkington AG, McKenna WJ, Mehta A, Pennell DJ, Leed PJ, Elliott PM. Gadolinium enhanced cardiovascular magnetic resonance in Anderson-Fabry disease. Evidence for a disease specific abnormality of the myocardial interstitium. Eur Heart J. 2003 Dec;24(23):2151-5. doi: 10.1016/j.ehj.2003.09.017. PMID 14643276
- [Background] Koeppe S, Neubauer H, Breunig F, Weidemann F, Wanner C, Sandstede J, Machann W, Hahn D, Kostler H, Beer M. MR-based analysis of regional cardiac function in relation to cellular integrity in Fabry disease. Int J Cardiol. 2012 Sep 20;160(1):53-8. doi: 10.1016/j.ijcard.2011.03.023. Epub 2011 Apr 3. PMID 21463907
- [Background] Kramer J, Niemann M, Stork S, Frantz S, Beer M, Ertl G, Wanner C, Weidemann F. Relation of burden of myocardial fibrosis to malignant ventricular arrhythmias and outcomes in Fabry disease. Am J Cardiol. 2014 Sep 15;114(6):895-900. doi: 10.1016/j.amjcard.2014.06.019. Epub 2014 Jul 2. PMID 25073565
- [Background] Kramer J, Niemann M, Liu D, Hu K, Machann W, Beer M, Wanner C, Ertl G, Weidemann F. Two-dimensional speckle tracking as a non-invasive tool for identification of myocardial fibrosis in Fabry disease. Eur Heart J. 2013 Jun;34(21):1587-96. doi: 10.1093/eurheartj/eht098. Epub 2013 Mar 21. PMID 23520186
- [Background] Bottomley PA, Foster TH, Argersinger RE, Pfeifer LM. A review of normal tissue hydrogen NMR relaxation times and relaxation mechanisms from 1-100 MHz: dependence on tissue type, NMR frequency, temperature, species, excision, and age. Med Phys. 1984 Jul-Aug;11(4):425-48. doi: 10.1118/1.595535. PMID 6482839
- [Background] Pica S, Sado DM, Maestrini V, Fontana M, White SK, Treibel T, Captur G, Anderson S, Piechnik SK, Robson MD, Lachmann RH, Murphy E, Mehta A, Hughes D, Kellman P, Elliott PM, Herrey AS, Moon JC. Reproducibility of native myocardial T1 mapping in the assessment of Fabry disease and its role in early detection of cardiac involvement by cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2014 Dec 5;16(1):99. doi: 10.1186/s12968-014-0099-4. PMID 25475749
- [Background] Thompson RB, Chow K, Khan A, Chan A, Shanks M, Paterson I, Oudit GY. T(1) mapping with cardiovascular MRI is highly sensitive for Fabry disease independent of hypertrophy and sex. Circ Cardiovasc Imaging. 2013 Sep;6(5):637-45. doi: 10.1161/CIRCIMAGING.113.000482. Epub 2013 Aug 6. PMID 23922004
- [Background] Pedrizzetti G, Claus P, Kilner PJ, Nagel E. Principles of cardiovascular magnetic resonance feature tracking and echocardiographic speckle tracking for informed clinical use. J Cardiovasc Magn Reson. 2016 Aug 26;18(1):51. doi: 10.1186/s12968-016-0269-7. PMID 27561421
- [Background] Tijsen AJ, Creemers EE, Moerland PD, de Windt LJ, van der Wal AC, Kok WE, Pinto YM. MiR423-5p as a circulating biomarker for heart failure. Circ Res. 2010 Apr 2;106(6):1035-9. doi: 10.1161/CIRCRESAHA.110.218297. Epub 2010 Feb 25. PMID 20185794
- [Background] Fichtlscherer S, De Rosa S, Fox H, Schwietz T, Fischer A, Liebetrau C, Weber M, Hamm CW, Roxe T, Muller-Ardogan M, Bonauer A, Zeiher AM, Dimmeler S. Circulating microRNAs in patients with coronary artery disease. Circ Res. 2010 Sep 3;107(5):677-84. doi: 10.1161/CIRCRESAHA.109.215566. Epub 2010 Jul 1. PMID 20595655
- [Background] Zampetaki A, Kiechl S, Drozdov I, Willeit P, Mayr U, Prokopi M, Mayr A, Weger S, Oberhollenzer F, Bonora E, Shah A, Willeit J, Mayr M. Plasma microRNA profiling reveals loss of endothelial miR-126 and other microRNAs in type 2 diabetes. Circ Res. 2010 Sep 17;107(6):810-7. doi: 10.1161/CIRCRESAHA.110.226357. Epub 2010 Jul 22. PMID 20651284
- [Background] Jansen F, Yang X, Proebsting S, Hoelscher M, Przybilla D, Baumann K, Schmitz T, Dolf A, Endl E, Franklin BS, Sinning JM, Vasa-Nicotera M, Nickenig G, Werner N. MicroRNA expression in circulating microvesicles predicts cardiovascular events in patients with coronary artery disease. J Am Heart Assoc. 2014 Oct 27;3(6):e001249. doi: 10.1161/JAHA.114.001249. PMID 25349183
- [Background] Goren Y, Kushnir M, Zafrir B, Tabak S, Lewis BS, Amir O. Serum levels of microRNAs in patients with heart failure. Eur J Heart Fail. 2012 Feb;14(2):147-54. doi: 10.1093/eurjhf/hfr155. Epub 2011 Nov 25. PMID 22120965
- [Background] Mignani R, Pieruzzi F, Berri F, Burlina A, Chinea B, Gallieni M, Pieroni M, Salviati A, Spada M. FAbry STabilization indEX (FASTEX): an innovative tool for the assessment of clinical stabilization in Fabry disease. Clin Kidney J. 2016 Oct;9(5):739-47. doi: 10.1093/ckj/sfw082. Epub 2016 Sep 9. PMID 27679722
- [Background] Cammarata G, Scalia S, Colomba P, Zizzo C, Pisani A, Riccio E, Montalbano M, Alessandro R, Giordano A, Duro G. A pilot study of circulating microRNAs as potential biomarkers of Fabry disease. Oncotarget. 2018 Jun 8;9(44):27333-27345. doi: 10.18632/oncotarget.25542. eCollection 2018 Jun 8. PMID 29937989
- [Background] Baig S, Edward NC, Kotecha D, Liu B, Nordin S, Kozor R, Moon JC, Geberhiwot T, Steeds RP. Ventricular arrhythmia and sudden cardiac death in Fabry disease: a systematic review of risk factors in clinical practice. Europace. 2018 Sep 1;20(FI2):f153-f161. doi: 10.1093/europace/eux261. PMID 29045633
- [Background] Nordin S, Kozor R, Baig S, Abdel-Gadir A, Medina-Menacho K, Rosmini S, Captur G, Tchan M, Geberhiwot T, Murphy E, Lachmann R, Ramaswami U, Edwards NC, Hughes D, Steeds RP, Moon JC. Cardiac Phenotype of Prehypertrophic Fabry Disease. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007168. doi: 10.1161/CIRCIMAGING.117.007168. PMID 29853467
- [Background] Nordin S, Kozor R, Medina-Menacho K, Abdel-Gadir A, Baig S, Sado DM, Lobascio I, Murphy E, Lachmann RH, Mehta A, Edwards NC, Ramaswami U, Steeds RP, Hughes D, Moon JC. Proposed Stages of Myocardial Phenotype Development in Fabry Disease. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 2):1673-1683. doi: 10.1016/j.jcmg.2018.03.020. Epub 2018 May 16. PMID 29778854
- [Derived] Camporeale A, Bandera F, Pieroni M, Pieruzzi F, Spada M, Bersano A, Econimo L, Lanzillo C, Rubino M, Mignani R, Motta I, Olivotto I, Tanini I, Valaperta R, Chow K, Baroni I, Boveri S, Graziani F, Pica S, Tondi L, Guazzi M, Lombardi M. Effect of Migalastat on cArdiac InvOlvement in FabRry DiseAse: MAIORA study. J Med Genet. 2023 Sep;60(9):850-858. doi: 10.1136/jmg-2022-108768. Epub 2023 Jan 20. PMID 36669872